CLINICAL TRIAL: NCT06259760
Title: Incidence and Risk Factors Analysis of Acute Kidney Injury (AKI) After Intentional Hypotensive Anesthesia in Orthognathic Surgery Patients Following Enhanced Recovery After Surgery (ERAS) Guidelines
Brief Title: AKI Risk Factors Analysis After Intentional Hypotensive Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-E(I)-20240015
Record Dates: First submitted 2024-02-07; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Acute Kidney Injury (Nontraumatic); Hypotension Drug-Induced
Keywords: Acute Kidney Injury; orthognathic surgery; general anesthesia; prospective analysis; intentional hypotension
MeSH Terms: conditions — Acute Kidney Injury; Hypotension | interventions — Nitroglycerin; Labetalol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Nitroglycerin — during surgery, the patient received nitroglycerin infusion or nitroglycerin with labetalol to decrease blood pressure and to decrease blood loss. During the procedures and management, patients were executed of continuously monitoring of arterial blood pressure, hemodynamic changes such as cardiac output, stroke volume variation, peripheral oxygen saturation, and cerebral oximeter.
  Other Names: labetalol

SUMMARY:
This project investigates intentionally hypotensive management such as NTG (nitroglycerin) or NTG+Trandate during general anesthesia in patients undergoing orthognathic surgery. Throughout the entire surgical procedure, blood biochemical and urine monitoring will be conducted. Serum creatinine (Cr) levels, urine analysis, and perioperative monitoring will be utilized as indicators for assessing renal function during the surgery. The objective is to assess its potential renal injury and identify early risk factors for acute kidney injury (AKI). Timely recognition of these factors will allow for the implementation of appropriate intervention strategies, aiding in the prevention of postoperative acute kidney injury. This approach contributes to achieving the goals of Enhanced Recovery After Surgery (ERAS) for surgical patients, promoting faster postoperative recovery.

DETAILED DESCRIPTION:
Orthognathic surgery is currently a common procedure in oral and maxillofacial surgery. The facial region is composed of a complex and dense vascular network, requiring precise, accurate, and delicate surgical techniques on both hard and soft tissues. During intraoral procedures, the surgical field may be limited, making the management of surgical bleeding challenging. Controlled hypotension or hypotensive anesthesia is often employed during major maxillofacial surgeries to optimize conditions. Lowering blood pressure is advantageous as it helps reduce overall blood loss and improves the surgeon's visibility. Therefore, maintaining stable blood pressure within the ideal range during the surgical process is a critical anesthesia objective.

This research emphasizes the prevention of acute kidney injury (AKI) in patients undergoing orthognathic surgery with intentional hypotension during general anesthesia. The goal is to detect the potential renal damage at an early stages, before a significant decline in kidney function occurs, thereby reducing the likelihood of acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* America society anesthesiologist classification class I to II patients undergoing oro-maxillo-facial surgery
* unlimited mouth opening

Exclusion Criteria:

* patients with arthritis with limited mouth opening
* persistent liver dysfunction
* chronic renal insufficiency
* body mass index ≧35 kg/m2.
* past history of malignant hyperthermia or personal or family history
* diabetes with insulin treatment
* essential hypertension without controlled

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients without obviously systemic diseases who presentation of abnormal oro-maxillofacial anatomy needs to be corrected.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
urine biomarkers assessment, urine output, and blood Creatinine from participants undergoing Orthognathic surgery. | intraoperative and postoperative stages, assessed up to 24 hours
  Record blood and urine biomarkers, and urine output after operation
permitted hypotension during surgery | intraoperative 2-6 hours
  assess intraoperative blood loss and the dosage of hypotensive medications to decrease intra-operative bleeding as patient undergoing oromaxillofacial surgery, intentional hypotension is allowed. however, adequate depth of anesthesia, proper cardiac output, respiratory parameters, temperatures should be monitored
consumption of inhaled and intravenous anesthetics | intraoperative 2-6 hours
  to maintain adequate depth of anesthesia during intentional hypotension, consumptions of inhaled and intravenous anesthetics are calculated

SECONDARY OUTCOMES:
time to successfully extubate the nasotracheal tube after anesthesia | from the end of surgery to the post-anesthesia care, assessed up to one hour
  early extubation allowable
safely discharged from post-anesthesia care unit (postoperative recovery room) | 2 hours
  as calculating the time from patient is delivered to postoperative recovery room to be safely discharged from recovery room by using the aldrete scores (activities level, respiration, circulation, conscious level, oxygenation) full back to pre-operative level or ten scores.
side effects and adverse events | intraoperative and postoperative stages, assessed up to 48 hours
  records any abnormal surgical or anesthesia related findings during this admission

CONTACTS AND LOCATIONS:
Overall Officials: Kuang-I Cheng, Phd, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Sanmin Dist, Taiwan